CLINICAL TRIAL: NCT02387619
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Rosuvastatin and Telmisartan/Amlodipine in Healthy Male Volunteers
Brief Title: The Pharmacokinetic Drug Interaction Between Rosuvastatin and Telmisartan/Amlodipine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1401-P1-DI
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Rosuvastatin Calcium; telmisartan amlodipine combination; Telmisartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 of part 1 (Experimental): Rosuvastatin and Telmisartan/Amlodipine: Rosuvastatin 20mg 1T during the period 1 and Rosuvastatin 20mg 1T and Telmisartan/Amlodipine 40/5mg 2T during the period 2
  Interventions: Drug: Rosuvastatin; Drug: Rosuvastatin and Telmisartan/Amlodipine
- Group 2 of part 1 (Experimental): Rosuvastatin and Telmisartan/Amlodipine: Rosuvastatin 20mg 1T, Telmisartan/Amlodipine 40/5mg 2T during the period 1 and Rosuvastatin 20mg 1T during the period 2
  Interventions: Drug: Telmisartan/Amlodipine; Drug: Rosuvastatin and Telmisartan/Amlodipine
- Group 1 of part 2 (Experimental): Rosuvastatin and Telmisartan/Amlodipine: Telmisartan/Amlodipine 40/5mg 2T during the period 1 and Rosuvastatin 20mg 1T, Telmisartan/Amlodipine 40/5mg 2T during the period 2
  Interventions: Drug: Rosuvastatin; Drug: Rosuvastatin and Telmisartan/Amlodipine
- Group 2 of part 2 (Experimental): Rosuvastatin and Telmisartan/Amlodipine: Rosuvastatin 20mg 1T, Telmisartan/Amlodipine 40/5mg 2T during the period 1 and Telmisartan/Amlodipine 40/5mg 2T during the period 2
  Interventions: Drug: Telmisartan/Amlodipine; Drug: Rosuvastatin and Telmisartan/Amlodipine

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin and Telmisartan/Amlodipine: Rosuvastatin once daily for 9 days
  Other Names: Crestor
  Arms: Group 1 of part 1; Group 1 of part 2
Drug: Telmisartan/Amlodipine — Rosuvastatin and Telmisartan/Amlodipine: Telmisartan/Amlodipine once daily for 9 days
  Other Names: Twynsta
  Arms: Group 2 of part 1; Group 2 of part 2
Drug: Rosuvastatin and Telmisartan/Amlodipine — Rosuvastatin and Telmisartan/Amlodipine: Rosuvastatin and Telmisartan/Amlodipine once daily for 9days
  Other Names: Crestor and Twynsta

SUMMARY:
A randomized, open-label, multiple-dose, crossover study to investigate the pharmacokinetic drug interaction between rosuvastatin and telmisartan/amlodipine in healthy male volunteers

DETAILED DESCRIPTION:
A randomized, open-label, 2-treatment, 2-sequence, 2-period, multiple-dose, crossover design

ELIGIBILITY:
Inclusion Criteria:

* 19~55 years healthy male
* Body weight is over 55kg, The result of Body Mass Index(BMI) is not less than 18 kg/m2 , no more than 27 kg/m2
* Subjects who agree to keep contraceptive methods during the clinical trial.

Exclusion Criteria:

* Subjects who are allergic to investigational drug.
* Subjects who have a medical history which can affect the clinical trial.
* Hypertension(Systolic BP ≥ 150mmHG or Diastolic BP ≥ 100mmHg), Hypotension(Systolic BP ≤ 100mmHg or Diastolic BP ≤ 65mmHg)
* Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss , Cmax, ss of Rosuvastatin and Telmisartan, Amlodipine | 72hours, 144hours

SECONDARY OUTCOMES:
AUClast,ss of Rosuvastatin | 72hours
AUCinf,ss of Rosuvastatin | 72hours
Tmax,ss of Rosuvastatin | 72hours
t1/2 of Rosuvastatin | 72hours
AUClast,ss of Telmisartan, Amlodipine | 144hours
AUCinf,ss of Telmisartan, Amlodipine | 144hours
Tmax,ss of Telmisartan, Amlodipine | 144hours
t1/2 of Telmisartan, Amlodipine | 144hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsoo Park, MD, Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Health System, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No